CLINICAL TRIAL: NCT04580277
Title: A Single Center Open-Label Prospective Study Of Oral Tofacitinib In Patients With Chronic Pouchitis
Brief Title: Tofacitinib For Treatment Of Chronic Pouchitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gil Melmed, Professor of Medicine, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000693
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Pouchitis; Ileal Pouchitis; Ileal Pouch
Keywords: chronic pouchitis; tofacitinib; antibiotic-refractory pouchitis; antibiotic-dependent pouchitis
MeSH Terms: conditions — Pouchitis | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic pouchitis (Experimental): This arm will include subjects with chronic pouchitis and will receive tofactinib 10 mg twice daily for 8 weeks
  Interventions: Drug: Tofacitinib 10 mg

INTERVENTIONS:
Drug: Tofacitinib 10 mg — Subjects in this arm will receive tofactinib 10 mg twice daily for 8 weeks

SUMMARY:
A phase 2 pilot study to evaluate the effectiveness of tofacitinib in subjects with chronic pouchitis

DETAILED DESCRIPTION:
The proposed study is a phase 2, open-label study of tofactinib in treatment of patients with chronic pouchitis. Subjects with chronic active pouchitis will be screened and recruited if they meet eligibility criteria. Eligible subjects will undergo baseline clinical evaluation, laboratory testing and a pouch endoscopy. They will then receive oral tofacitinib 10 mg twice daily for 8 weeks. Clinical and laboratory data will be collected at week 4 and week 8, and all subjects will undergo a end of treatment pouch endoscopy at 8 weeks. Clinical, laboratory and endoscopic data at 8 weeks will be compared to the baseline data to evaluate study outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ages 18 to 80
2. Subjects with a history of proctocolectomy with ileal pouch anal anastomosis (IPAA) for UC at least 6 months prior to screening.
3. Subjects with pouchitis that is chronic, defined by a mPDAI score ≥5 assessed as the average from 3 days immediately prior to the baseline study visit and a minimum endoscopic sub-score of 2 (outside the staple or suture line) with either (a) ≥ 3 recurrent episodes within 1 year prior to the screening treated with ≥2 weeks of antibiotic or other prescription therapy, (b) requiring maintenance antibiotic therapy taken continuously for ≥4 weeks immediately prior to the baseline study visit
4. Women of childbearing potential must have documentation of a negative pregnancy test at screening and must agree to use two highly effective methods of birth control during the study and for at least 1 month after completion of study drug dosing.

Exclusion Criteria:

1. Subjects with IPAA surgery done for Crohn's disease (CD) or familial adenomatous polyposis (FAP) indications.
2. Subjects with primary CD of pouch, isolated or predominant cuffitis or mechanical complications of the ileal pouch.
3. Subjects with prior exposure to tofacitinib.
4. Subjects with a diverting stoma.
5. Subjects with a prior history or risk factors for venous thromboembolism.
6. Subjects with active bacterial, parasitic, fungal, mycobacterial, or viral infection.
7. Subjects with a history of latent or active tuberculosis.
8. Subjects positive for hepatitis B virus (HBV) surface antigen, hepatitis B virus core antibody with a negative hepatitis B surface antibody or with detectable serum hepatitis B DNA.
9. Female subjects who are pregnant or lactating.
10. Female subjects of childbearing potential who are sexually active and do not agree to using two highly effective methods of contraception during the study period.
11. Subjects with clinically significant laboratory abnormalities at study screening.

    * Other eligibility criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven patients were screened and 6 met the eligibility criteria. One patient was ineligible due to an endoscopic PDAI subscore of 1 on screening pouchoscopy. Study recruitment was terminated prematurely due to COVID-19 pandemic-related recruitment challenges.
Groups:
- Chronic Active Pouchitis: This arm included subjects with chronic active pouchitis who recieved tofactinib 10 mg twice daily for 8 weeks
  Tofacitinib 10 mg: Subjects in this arm will receive tofactinib 10 mg twice daily for 8 weeks
Period: Overall Study
Arm/Group | Chronic Active Pouchitis
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: Years] | 23.5 [19 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Prior Biologic Use for Pouchitis [Count of Participants; unit: Participants] | 6
Indication for Colectomy [Count of Participants; unit: Participants]
  Active ulcerative colitis | 6
  Dysplasia/cancer | 0
Concomitant Medications [Count of Participants; unit: Participants] — Study subjects were allowed to remain on permitted concomitant medications provided the patient was on a stable dose for ≥2 weeks prior to starting tofactinib. Patients stayed on stable doses of these medications for the study duration of 8 weeks.
  Participants
    On Antibiotics | 4
    On Corticosteroids | 1
    On Immunomodulators | 0
    Other | 1
Extraintestinal Manifestations [Count of Participants; unit: Participants]
  Arthritis | 2
  Primary sclerosing cholangitis | 1
  Other | 0
  None | 3
Median Baseline mPDAI score [Median (Full Range); unit: PDAI score] — The modified PDAI (mPDAI), which can range from 0 to 12, is calculated from 2 separate 6-point scales assessing clinical symptoms and endoscopic findings. Patients are classified as either having pouchitis (PDAI score ≥5) or as not having pouchitis (PDAI score <5). Greater clinical scores and endoscopy scores correspond to worse disease severity."
  PDAI score | 8.8 [7 to 10]
Median Baseline Fecal Calprotectin [Median (Full Range); unit: mcg/g] | 217 [28 to 1340]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response/Remission
Description: The proportion of subjects with clinical response at 8 weeks, defined as ≥2-point decrease in modified pouchitis disease activity index (mPDAI) with at least 1-point decrease in endoscopic subscore compared to the baseline.The mPDAI is a 0- 18 point scale of pouchitis disease severity, with higher scores corresponding to worse disease severity.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
Participants | 4

2. Secondary Outcome: Number of Participants With Clinical Response
Description: The proportion of subjects with clinical remission at 8 weeks, defined as modified pouchitis disease activity index (mPDAI) <5.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
Participants | 4

3. Secondary Outcome: Number of Participants With Clinical Remission
Description: The proportion of subjects with clinical remission at 8 weeks, defined as a modified pouch disease activity index (mPDAI) score of <5 with a ≥2-point decrease from the baseline mPDAI score. The mPDAI is a 0- 18 point scale of pouchitis disease severity, with higher scores corresponding to worse disease severity.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
Participants | 3

4. Secondary Outcome: Change in mPDAI Score
Description: change in median mPDAI score at 8 weeks compared to baseline. The mPDAI (modified pouchitis disease activity index) is a 0- 18 point scale of pouchitis disease severity, with higher scores corresponding to worse disease severity.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
score on a scale | -4.5 [-8.33 to -4.34]

5. Secondary Outcome: Change in mPDAI Clinical Sub-score
Description: change in median clinical mPDAI sub-score at 8 weeks compared to baseline. The mPDAI (modified pouchitis disease activity index) is a 0- 18 point scale of pouchitis disease severity, with higher scores corresponding to worse disease severity.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
score on a scale | -1.7 [-2.33 to -1.34]

6. Secondary Outcome: Change in mPDAI Endoscopic Sub-score
Description: change in median endoscopic mPDAI sub-score at 8 weeks compared to baseline. The mPDAI (modified pouchitis disease activity index) is a 0- 18 point scale of pouchitis disease severity, with higher scores corresponding to worse disease severity.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
score on a scale | -2 [-6 to -1]

7. Secondary Outcome: Change in IBD-related Quality of Life
Description: CGQL is a quality of life questionnaire used in inflammatory bowel diseases that incorporates three domains - quality of life, quality of health and energy level. Each domain is scored from 0 (worst) to 10 (best)and a total score is calculated by dividing the cumulative score by 30. The CGQL score can range from 0 to 1. Change in quality of life as measured by the Cleveland Global Quality of Life score (CGQL) at 8 weeks compared to baseline.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Chronic Active Pouchitis
Number analyzed (Participants) | 6
score on a scale | 0.1 [0 to 0.3]

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored from the beginning of the study (week 0) up to 12 weeks (4 weeks after the completion of the study)
Arm/Group | Chronic Pouchitis
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Pouchitis (N=6)
Sepsis (Gastrointestinal disorders) | 1 (1) — Patient hospitalized with sepsis related to shigella infection after starting tofacitinib. This patient recovered completely, resumed tofacitinib after a 6-day treatment interruption and completed the 8-week study.
Pouchitis Flare/SMA (superior mesentery artery) syndrome (Gastrointestinal disorders) | 1 (1) — Event was unrelated to Investigational Drug. Participant recovered without sequelae.
Severe Malnutrition/failure to thrive secondary to SMA syndrome (Metabolism and nutrition disorders) | 1 (1) — Event was unrelated to Investigational Drug and participant recovered without sequelae.
worsening of superior mesenteric artery syndrome (Gastrointestinal disorders) | 1 (1) — Event outcome is ongoing and unrelated to Investigational Drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic Pouchitis (N=6)
Worsening of pouchitis disease symptoms (Gastrointestinal disorders) | 1 (1) — Event was moderate in severity and unrelated to Investigational Drug.
Flu-like symptom (General disorders) | 1 (1) — Event was mild in severity and unrelated to Investigational Drug. Participant recovered without sequelae.
COVID-19 test positive (General disorders) | 1 (1) — Event was mild in severity and unrelated to Investigational Drug. Patient recovered without sequelae.

LIMITATIONS AND CAVEATS:
Limitations of this study included a single center design, small sample size, and absence of a control arm. This study also lacked long-term follow-up data to assess durability of response to tofacitinib and its long-term safety in chronic pouchitis. This study also only included patients with chronic pouchitis and its findings may not be applicable to other chronic inflammatory pouch disorders. Study recruitment was terminated prematurely due to COVID-19 pandemic-related recruitment challenges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT04580277/Prot_SAP_001.pdf